CLINICAL TRIAL: NCT06926296
Title: Moral Injury in French Healthcare Workers
Acronym: MI-PRO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024-CHITS-019; 2024-a02449-38 (Other: ID-RCB number)
Record Dates: First submitted 2025-04-07; First posted 2025-04-13 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Moral Injury
Keywords: Moral injury; Burnout; Depression; Anxiety; Healthcare workers; Health services research
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Burnout, Psychological; Depression; Anxiety Disorders | interventions — Health Personnel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthcare workers (Other): All health professionals working in metropolitan France and the French overseas departments and territories
  Interventions: Other: Self-Questionnaires for Healthcare Workers

INTERVENTIONS:
Other: Self-Questionnaires for Healthcare Workers — Health workers will be invited to complete an online self-questionnaire.

SUMMARY:
Healthcare professionals are facing an escalating crisis, with burnout rates ranging between 40% and 60% and a growing intention to leave the profession, affecting one in five physicians and one in four nurses in the coming years. While current interventions focused on individual resilience, such as mindfulness, peer support, and workload management, have been promoted as solutions, they have failed to bring about systemic improvements. This raises the question of whether other factors, such as Moral Injury, play a key role in this crisis. Moral Injury is an emerging concept that highlights the profound misalignment between healthcare workers' professional values and the reality of their practice, often exacerbated by organizational and economic constraints.

The objective of this study is to describe the manifestations of Moral Injury among healthcare professionals in France. By establishing the first large-scale assessment of Moral Injury among healthcare professionals in France, this study aims to identify key organizational and personal risk factors contributing to this phenomenon. The use of Structural Equation Modeling will help build a robust theoretical model that clarifies the underlying mechanisms of Moral Injury and its interactions with broader health issues. The findings will support the development of targeted interventions focused on systemic organizational changes to improve healthcare workers' well-being and guide public health policies.

DETAILED DESCRIPTION:
Healthcare professionals are facing an escalating crisis, with burnout rates ranging between 40% and 60% and a growing intention to leave the profession, affecting one in five physicians and one in four nurses in the coming years. While current interventions focused on individual resilience, such as mindfulness, peer support, and workload management, have been promoted as solutions, they have failed to bring about systemic improvements. This raises the question of whether other factors, such as Moral Injury, play a key role in this crisis. Moral Injury is an emerging concept that highlights the profound misalignment between healthcare workers' professional values and the reality of their practice, often exacerbated by organizational and economic constraints.

The primary objective of this study is to describe the manifestations of Moral Injury among healthcare professionals in France. Secondary objectives include the psychometric validation of a French-language Moral Injury scale, the analysis of organizational and individual determinants of Moral Injury, and the structural modeling of underlying mechanisms.

This nationwide cross-sectional survey will be conducted electronically, reaching participants through healthcare institutions, professional societies, social networks, and a snowball dissemination strategy. Data collection will include standardized scales such as the Moral Injury Inventory for Healthcare Professionals, the Moral Injury Events Scale (MIES), the Maslach Burnout Inventory (MBI), and the EuroQol 5-Dimensions (EQ-5D) for quality of life, as well as ad hoc questions designed to explore additional systemic and professional challenges. A rigorous psychometric validation of the Moral Injury scale will be performed, followed by Structural Equation Modeling (SEM) to analyze the complex relationships between Moral Injury and other factors such as burnout, depression, and anxiety.

By establishing the first large-scale assessment of Moral Injury among healthcare professionals in France, this study aims to identify key organizational and personal risk factors contributing to this phenomenon. The use of Structural Equation Modeling will help build a robust theoretical model that clarifies the underlying mechanisms of Moral Injury and its interactions with broader health issues. The findings will support the development of targeted interventions focused on systemic organizational changes to improve healthcare workers' well-being and guide public health policies.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare workers

Exclusion Criteria:

* Absence of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3073 (Estimated)
Dates: Start 2025-11-19 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Moral Injury Inventory for Healthcare Professionals | One point : baseline
  An overall score out of 100 will be created for the inventory, where a high score indicates a high level of "Moral Injury"

SECONDARY OUTCOMES:
Moral Injury Events Scale | One point : baseline
  Minimum score = 11, Maximum score = 66 Higher average scores indicate greater intensity of experience
Maslach Burnout Inventory | One point : baseline
  3 scores calculated in this inventory Burnout : minimum score = 0, maximum score = 63, Higher average scores indicate greater intensity of burnout Depersonalization : minimum score = 0, maximum score = 35, Higher average scores indicate greater intensity of depersonalization Personal fulfillment : minimum score = 0, maximum score = 56, Higher average scores indicate greater intensity of personal fulfillment
EuroQol 5-Dimensions (EQ-5D) | One point : baseline
  Scores range from -0.59 to 1, where 1 is the best possible health status.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent BOYER, Pr, Study Director — CEReSS
Locations (1):
- Centre Hospitalier Intercommunal Toulon-La Seyne sur Mer, Toulon, Var, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boyer L, Fond G, Tran B, Llorca PM, Duclos A. The hidden crisis: Moral injury among French healthcare workers. J Epidemiol Popul Health. 2024 Dec;72(6):202780. doi: 10.1016/j.jeph.2024.202780. Epub 2024 Oct 19. PMID 39427511
- [Background] Dean W, Morris D, Llorca PM, Talbot SG, Fond G, Duclos A, Boyer L. Moral Injury and the Global Health Workforce Crisis - Insights from an International Partnership. N Engl J Med. 2024 Sep 5;391(9):782-785. doi: 10.1056/NEJMp2402833. Epub 2024 Aug 31. No abstract available. PMID 39216090